CLINICAL TRIAL: NCT01550458
Title: A Study of the Pharmacokinetic and Safety Profile of QID Dosing of Mibefradil in Normal Human Volunteers
Brief Title: Safety Study of Mibefradil When Given Four Times a Day in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cavion, Inc. (Industry)
Collaborators: Celerion (Industry); Dana-Farber Cancer Institute (Other); LifeWatch Services, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cavion (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAU-2011-01
Record Dates: First submitted 2012-02-29; First posted 2012-03-12 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Clinical Trial, Phase I; Human Volunteers; Healthy Volunteers; mibefradil; Posicor®
MeSH Terms: interventions — Mibefradil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mibefradil (Experimental)
  Interventions: Drug: mibefradil
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: mibefradil — 25 mg tablets for oral administration given for 7 days at a total daily dose beginning at 100 mg per day divided into four doses. Doses will be incremented in successive cohorts by 25 mg/day up to 400 mg/day.
  Other Names: Posicor®; mibefradil dihyrdochloride; RO 40-5967
  Arms: Mibefradil
Other: Placebo — 1 out of 6 patients per cohort will receive placebo tablets identical in appearance and number to the active mibefradil arm.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The objective of the study is to determine the safety and pharmacokinetics of a 7 day course of oral mibefradil given four times a day in healthy volunteers. This is a dose escalation study in which the total daily dose of mibefradil will be increased with each cohort.

DETAILED DESCRIPTION:
This study will establish the safety, detailed pharmacokinetics, and, possibly, maximum tolerated dose (MTD) of ascending doses of mibefradil administered four times a day (QID) in healthy volunteers. The knowledge gained will then guide the details of a study of Interlaced Therapy™ in patients with recurrent High Grade Glioma (HGG). Non-clinical studies are currently on-going in the efficacy of Interlaced Therapy™ in ovarian cancer, pancreatic cancer, and intracranial malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy volunteers aged 19 to 55 years, male or female, and willing and able to sign informed consent;
2. Females must have a negative pregnancy test at screening and be practicing a suitable method of birth control so that, in the opinion of the Investigator, they will not become pregnant during the course of the study, or females can be postmenopausal (no menstrual period for one year) or surgically sterilized. Females must either be sexually inactive (abstinent) for 14 days prior to Screening and remain so through 30 days following the final dosing of the study drug or have been using one of the following acceptable methods of birth control for the times specified:

   * Barrier method (condom or diaphragm) with spermicidal for at least 14 days prior to Screening through Day -1 through 30 days following the final dosing of the study drug;
   * Surgical sterilization (vasectomy) of partner at least 6 months prior to Day -1; or
   * Females of non-childbearing potential have undergone one of the following sterilization procedures at least 6 months prior to Day -1: bilateral tubal ligation, hysterectomy, hysterectomy with unilateral or bilateral oophorectomy, or bilateral oophorectomy.
3. Male subjects must continue to use their approved contraceptive method for 60 days after participating in the study.
4. Has a body mass index (BMI) between 18.0 and 32.0 kg/m², inclusive; and
5. Have no acute illnesses or chronic health issues that require medication.

Exclusion Criteria:

1. History of investigational drug use within 30 days of this study;
2. Subject has a clinically significant disorder that, in the opinion of the Investigator, could result in the subject's inability to understand and comply with the requirements of the study;
3. History of hypertension, treated or untreated, or screening BP >140 mm Hg systolic or >90 mm Hg diastolic;
4. Currently or within the last 14 days taking any medications (prescription, nonprescription, or herbal or Chinese remedies) including oral contraceptives and hormone replacement therapy;
5. Subject has a history of impaired hepatic function that, in the Investigator's opinion, contraindicates participation in this study; or the subject has any other abnormal laboratory value of clinical significance for this study in the Investigators opinion;
6. Current smoker (more than 10 cigarettes/day) for 6 months;
7. Subject has a creatinine clearance (CLcr) of less than 70 mL/min as calculated by the

   Cockroft-Gault equation:

   CLcr = ((140 - age) x body mass x [0.85 if female]) / (72 x creatinine)

   where age is given in years, body mass is given in kg, and creatinine is given in mg/dL;
8. Subject has a history, signs, or symptoms of ischemic cardiac, cerebrovascular, or peripheral vascular syndromes or other significant underlying cardiovascular disease that are clinically significant in the Investigator's opinion. This includes any known cardiac rhythm disorder or ECG abnormality;
9. Subject, in the Investigator's opinion, is likely to have unrecognized cardiovascular disease, based on history or the presence of risk factors;
10. Subject is currently taking or had taken in the previous 14 days, herbal preparations containing St. John's Wort (Hypericum perforatum);
11. Subject has a history of allergic reactions to calcium channel antagonists;
12. Females who are pregnant, actively trying to become pregnant, or lactating. Females must be practicing a suitable method of birth control (adequate barrier method of birth control; abstinence) so that, in the opinion of the Investigator, they will not become pregnant during the course of the study, or females can be postmenopausal (no menstrual period for one year) or surgically sterilized;
13. Subject had a recent history (in the past 3 months) suggestive of evidence of alcohol or drug abuse or dependence, or has any unaccounted-for drug or alcohol in the original drug screen (tested positive);
14. Allergy to latex or rubber;
15. Hemoglobin under laboratory lower limit of normal; or
16. Significant blood loss of 500 mL or greater or blood donation within 56 days prior to Day 1. Subjects cannot donate plasma within 5 days prior to Day 1.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06-24 (Actual); Study Completion 2012-06-24 (Actual)

PRIMARY OUTCOMES:
Determine the safety of a 7-day course of oral mibefradil in four divided daily doses in normal healthy volunteers. | 7 days
  Safety will be assessed by clinical laboratory tests, physical examinations, vital sign measurements, continuous, real time, 3-lead ECG monitoring, concomitant medication documentation and adverse event monitoring.

SECONDARY OUTCOMES:
Steady State Cmax of Mibefradil | daily for 7 days
  Pharmacokinetics assessments will include the determination of plasma concentrations of mibefradil and its major metabolite. Blood samples will be drawn on Day 1: pre-dose 1, 30 minutes, 1 hr, 2 hr, 3 hr, 4 hr, pre-dose 2, pre-dose 3, pre-dose 4; Day 2: pre-dose 1, pre-dose 3; Day 3: pre-dose 1, pre-dose 3; Day 4: pre-dose 1, 30 minutes, 1 hr, 2 hr, 3 hr, 4 hr, pre-dose 2, pre-dose 3; Day 5: pre-dose 1, pre-dose 3; Day 6: pre-dose 1, pre-dose 3; and Day 7: pre-dose 1, pre-dose 3, pre-dose 4, 30 minutes, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 7 hr, 9 hr after dosing.
Half Life of Mibefradil | daily for 7 days
  Pharmacokinetics assessments will include the determination of plasma concentrations of mibefradil and its major metabolite. Blood samples will be drawn on Day 1: pre-dose 1, 30 minutes, 1 hr, 2 hr, 3 hr, 4 hr, pre-dose 2, pre-dose 3, pre-dose 4; Day 2: pre-dose 1, pre-dose 3; Day 3: pre-dose 1, pre-dose 3; Day 4: pre-dose 1, 30 minutes, 1 hr, 2 hr, 3 hr, 4 hr, pre-dose 2, pre-dose 3; Day 5: pre-dose 1, pre-dose 3; Day 6: pre-dose 1, pre-dose 3; and Day 7: pre-dose 1, pre-dose 3, pre-dose 4, 30 minutes, 1 hr, 2 hr, 3 hr, 4 hr, 5 hr, 7 hr, 9 hr after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States